CLINICAL TRIAL: NCT01192984
Title: Phase II Study of KW-0761 in Subjects With CCR4-positive Peripheral T/NK-cell Lymphoma
Brief Title: Study of KW-0761 in Subjects With CCR4-positive Peripheral T/NK-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 0761-004
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Peripheral T/NK-cell Lymphoma
MeSH Terms: interventions — mogamulizumab

ARMS (1):
- KW-0761 (Experimental)
  Interventions: Biological: KW-0761

INTERVENTIONS:
Biological: KW-0761 — Intravenously 8 times at 1-week intervals

SUMMARY:
The purpose of this study is to evaluate the efficacy of KW-0761 intravenously administered eight times at one-week intervals in patients with CCR4-positive peripheral T/NK-cell lymphoma. The primary objective is to assess the antitumor effect in terms of best overall response, while the secondary objectives are to assess the antitumor effect in terms of best response by disease lesion, to assess the progression-free survival and to assess the overall survival. The safety and pharmacokinetic profiles of KW-0761 will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with hematologically or pathohistologically diagnosed peripheral T/NK-cell lymphoma
* Subjects who have been positive for CCR4
* Subjects who received one or more chemotherapy regimens
* Subjects who relapse after achieving complete response, uncertain complete response or partial response by the last chemotherapy
* Subjects who have an interval of 4 weeks or more between the last day of the prior therapy and the scheduled day of the first KW-0761 treatment
* Subjects with nodal lesions, extranodal lesions and/or cutaneous lesions
* Subjects who have a performance status of 0 to 2
* Subjects who are negative for HBs antigen and reported as "not detected" for HBV-DNA
* Subjects who are negative for anti-HCV antibody
* Subjects who have normal function of the major organs
* Subjects who have given written voluntary informed consent to participate in the study

Exclusion Criteria:

* Subjects who underwent transplant therapy such as hematopoietic stem-cell transplantation (Subjects who underwent autologous hematopoietic stem-cell transplantation following chemotherapy will not be excluded)
* Subjects who are known carriers of HIV
* Subjects who have active multiple cancer
* Subjects who have a history of allergic reactions to therapeutic antibodies
* Subjects requiring continuous systemic treatment with steroid
* Subjects who require emergency radiotherapy for treating the symptoms caused by bulky masses at enrollment or who may require such radiotherapy after the start of the study
* Subjects who are pregnant, lactating or of childbearing potential, or who are planning to have children

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Antitumor effect (best overall response)

SECONDARY OUTCOMES:
Antitumor effect (best response by disease lesion), progression-free survival and overall survival
Adverse events and anti-KW-0761 antibody levels
Plasma KW-0761 concentrations and pharmacokinetic parameters

CONTACTS AND LOCATIONS:
Locations (15):
- Japan (15):
  - Kyushu University Hospital, Fukuoka
  - National Kyushu Cancer Center, Fukuoka
  - Tokai University Hospital, Isehara
  - Imamura Bun-in Hospital, Kagoshima
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Nagasaki University Hospital, Nagasaki
  - Aichi Cancer Center Hospital, Nagoya
  - Nagoya City University Hospital, Nagoya
  - Nagoya Daini Red Cross Hospital,, Nagoya
  - Okayama University Hospital, Okayama
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Cancer Institute Hospital, Tokyo
  - National Cancer Center Hospital, Tokyo
  - Mie University Hospital, Tsu

REFERENCES:
- [Derived] Ogura M, Ishida T, Hatake K, Taniwaki M, Ando K, Tobinai K, Fujimoto K, Yamamoto K, Miyamoto T, Uike N, Tanimoto M, Tsukasaki K, Ishizawa K, Suzumiya J, Inagaki H, Tamura K, Akinaga S, Tomonaga M, Ueda R. Multicenter phase II study of mogamulizumab (KW-0761), a defucosylated anti-cc chemokine receptor 4 antibody, in patients with relapsed peripheral T-cell lymphoma and cutaneous T-cell lymphoma. J Clin Oncol. 2014 Apr 10;32(11):1157-63. doi: 10.1200/JCO.2013.52.0924. Epub 2014 Mar 10. PMID 24616310